CLINICAL TRIAL: NCT06508762
Title: A Phase 1, Open-label, Randomized, Crossover Study to Evaluate the Relative Bioavailability and Food Effect of a New Tablet Formulation of VX-993 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability and Food Effect of a New Tablet Formulation of VX-993
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX24-993-005
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-993 (Experimental): Participants will be randomized to receive VX-993 in 1 of 6 treatment sequences with 3 dosing periods to assess the relative bioavailability of two VX-993 formulations and the effect of food on the pharmacokinetics of VX-993.
  Interventions: Drug: VX-993

INTERVENTIONS:
Drug: VX-993 — Tablet and Suspension for Oral Administration.

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (PK), safety, and tolerability of VX-993 in healthy adult participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2), inclusive
* A total body weight of more than (>) 50 kg
* Nonsmoker or ex-smoker for at least 3 months before first dose of the study drug

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption, distribution, metabolism, or excretion

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-993 | From Day 1 up to Day 28
Area Under the Concentration Versus Time Curve for the Last Measurable Concentration (AUClast) of VX-993 | From Day 1 up to Day 28
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-993 | From Day 1 up to Day 28

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-993 Metabolite | From Day 1 up to Day 28
Area Under the Concentration Versus Time Curve for the Last Measurable Concentration (AUClast) of VX-993 Metabolite | From Day 1 up to Day 28
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-993 Metabolite | From Day 1 up to Day 28
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing